CLINICAL TRIAL: NCT04691804
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Study of Fuzuloparib Combined With Abiraterone Acetate and Prednisone (AA-P) Versus Placebo Combined With AA-P as First-Line Treatment in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR3162-III-305
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer (mCRPC)
MeSH Terms: interventions — Abiraterone Acetate; Prednisone; fluzoparib

STUDY DESIGN:
Intervention Model Description: Fuzuloparib Combined with Abiraterone Acetate and Prednisone (AA-P) versus Placebo Combined with AA-P
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group A (Experimental): Fuzuloparib plus AA-P
  Interventions: Drug: Fuzuloparib , Abiraterone acetate and Prednisone
- Treatment group B (Placebo Comparator): Fuzuloparib Placebo plus AA-P
  Interventions: Drug: Fuzuloparib Placebo， Abiraterone acetate and Prednisone

INTERVENTIONS:
Drug: Fuzuloparib , Abiraterone acetate and Prednisone — 1. Fuzuloparib capsules (strength: 50 mg),150mg, Bid,po
  2. Abiraterone acetate tablets (strength: 250 mg) 1000mg Qd,po
  3. Prednisone tablets (strength: 5 mg) 5mg, Bid po
  Other Names: SHR3162
  Arms: Treatment group A
Drug: Fuzuloparib Placebo， Abiraterone acetate and Prednisone — 1. Fuzuloparib capsules Placebo (strength: 50 mg),150mg, Bid,po
  2. Abiraterone acetate tablets (strength: 250 mg)1000mg Qd,po
  3. Prednisone tablets (strength: 5 mg)5mg, Bid po
  Arms: Treatment group B

SUMMARY:
To evaluate whether Fuzuloparib plus AA-P is superior to placebo plus AA-P as first-line treatment by assessment of radiographic progression-free survival (rPFS) in mCRPC subjects unselected for deoxyribonucleic acid (DNA) damage repair deficiencies (DRD) status (Cohort 1) to evaluate whether Fuzuloparib plus AA-P is superior to placebo plus AA-P as first-line treatment by assessment of rPFS in mCRPC subjects harboring DRD (Cohort 2).

ELIGIBILITY:
Inclusion Criteria

1. Able and willing to provide a written informed consent
2. A score of 0 to 1 for ECOG performance status
3. Age of ≥ 18 years old
4. Prostate adenocarcinoma confirmed
5. Disease progression of metastatic prostate cancer while the subject was on androgen deprivation therapy.
6. The functional level of the organs must meet the requirements
7. Blood and tumor tissue samples are provided during screening to determine the DRD status

Exclusion Criteria

1. Prior treatment with any PARP inhibitor
2. Have received any systemic anti-tumor treatment during the mCRPC stage or non-metastatic CRPC stage
3. Have used any CYP3A4 inducers or inhibitors within 14 days prior to the first dose
4. Plan to receive any other anti-tumor treatment
5. Presence of radiologically confirmed tumor lesions in the brain
6. Contraindications to the use of Prednisone
7. History of uncontrolled pituitary or adrenal dysfunction
8. Uncontrolled hypertension
9. Presence of active heart diseases
10. Human immunodeficiency virus-positive
11. Presence of dysphagia, chronic diarrhea, intestinal obstruction, or other factors affecting drug intake and absorption
12. Active HBV or HCV infection
13. Presence of concomitant diseases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rPFS by blinded independent central review (BICR) using RESIST1.1 and PCWG3 | up to 3 years
  progression-free survival

SECONDARY OUTCOMES:
OS | up to 4 years
  time from randomization to death due to any cause
ORR | up to 3 years
  The percentage of subjects with measureable disease at baseline who achieved a complete or partial response in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
Time to PSA progression | up to 3 years
  Time from randomisation to the first time of PSA progression according to the criterion of PCGW3
Time to skeletal-related events | up to 4 years
  Time from randomisation to the first occurrence of a fracture or treatment for the fracture. The skeletal-related event is defined as the occurrence of either pathological or clinical fracture, spinal cord compression, bone-related radiotherapy or surgery.

CONTACTS AND LOCATIONS:
Locations (147):
- United States (17):
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Urological Associates of Southern Arizona PC, Tucson, Arizona
  - Desert Hematology Oncology Medical Group Inc, Rancho Mirage, California
  - San Bernardino Urological Associates Medical Group, San Bernardino, California
  - UF College of Medicine - Jacksonville, Jacksonville, Florida
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - VA Maryland Health Care System, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - GU Research Network LLC, Omaha, Nebraska
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - Center for Onology and Blood Disorders, Houston, Texas
- Australia (10):
  - Bendigo Health, Bendigo
  - Concord Repatriation General Hospital, Concord
  - St Vincents Hospital Melbourne, Fitzroy
  - Gosford Hospital, Gosford
  - Ashford Cancer Centre Research, Kurralta Park
  - The Alfred Hospital, Melbourne
  - Western Health, St Albans
  - Macquarie University, Sydney
  - Riverina Cancer Care Centre, Wagga Wagga
  - Sydney Adventist Hospital, Wahroonga
- Belgium (3):
  - UZ Gent, Ghent
  - Centre Hospitalier de Jolimont, Haine-Saint-Paul
  - AZ Groeninge, Kortrijk
- China (56):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Beijing cancer hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Hospital, Beijing
  - Cancer hospital Chinese academy of medical science, Beijing
  - Hunan Cancer Hospital, Changsha
  - XiangYa hospital central south university, Changsha
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - The First affiliatared hospital of Fujian medical university, Fuzhou
  - Cancer Center, Sun Yat-sen University, Guangzhou
  - Sun Yet-Sen Memorial Hospital,Sun Yet-Sen University, Guangzhou
  - Affiliated Hospital of Guizhou Medical University, Guiyang
  - Guizhou Cancer Hospital, Guiyang
  - The First Affiliated Hospital，ZheJiang University School of Medicine, Hangzhou
  - ZheJiang Provincial People's Hospital, Hangzhou
  - Urology Ward 2，Harbin Medical University Cancer Hospital, Ha’erbin
  - Anhui Provincial Hospital, Hefei
  - The First Affiliated Hospital Of Anhui Medical University, Hefei
  - The Second Hospital Of Anhui Medical University, Hefei
  - The First Hospital of Jiaxing, Jiaxing
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Provincial Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University-DepartmentDepartment of Urology, Nanchang
  - JiangSu Cancer Hospital, Nanjing
  - Jiangsu Province Hospitall, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - The first affiliated hospital of guangxi medical university, Nanjing
  - ZhongDa hospital southeast university, Nanjing
  - Qingdao Municipal Hospital, Qingdao
  - Changhai Hospital of Shanghai-Department of Urology, Shanghai
  - Shanghai Tenth People's Hospital-Department of Urology, Shanghai
  - The Urology Surgery department of Zhongshan Hospital, Shanghai
  - Liaoning Cancer Hospital, Shenyang
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - First Hospital of Shanxi Medical University, Taiyuan
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - The Second Hospital Of TianJin medical University, Tianjin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The Affiliated Tumor Hospital of Xinjiang Medical University-Department of Urology, Ürümqi
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital of Tongji Medical College,Huazhong University of Science and Technology, Wuhan
  - Union Hospital of Tongji Medical College,Huazhong University of Science and Technology, Wuhan
  - Wuxi People's Hospital-Department of Urinary Surgery, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Northern Jiangsu People's Hospital, Yangzhou
  - Henan Cancer Hospital, Zhengzhou
  - Henan Provincial People's Hospital, Zhengzhou
- Czechia (2):
  - Nemocnice Novy Jicin a.s., Nový Jičín
  - Thomayerova Nemocnice, Prague
- France (10):
  - Centre Hospitalier Departemental Vendee CHD, La Roche-sur-Yon
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Universitaire de Nimes, Institut de Cancerologie du Gard, Nîmes
  - Hopital Europeen George Pompidou, Paris
  - Hopital Lyon Sud, Pierre-Bénite
  - Centre Eugenie Marquis, Rennes
  - Centre de Lutte Contre le Cancer (CLCC) - Institut de Cancerologie de l'Ouest (ICO) - Rene Gauducheau, Saint-Herblain
  - Strasbourg Oncologie Liberale- Clinique Sainte Anne, Strasbourg
  - Institut Univ du Cancer de Toulouse-Oncopole, Toulouse
- Hungary (5):
  - National Institute of Oncology, Budapest
  - Semmelweis Egyetem, Budapest
  - Bekes Megyei Kozponti Korhaz, Gyula
  - BKMK Hospital, Kecskemét
  - Szent Borbala Korhaz, Tatabánya
- Poland (8):
  - Szpitale Pomorskie Sp.zo.o, Gdynia
  - Regionalny Szpital Specjalistyczny im.dr. Wladyslawa Bieganskiego, Grudziądz
  - Clinical Research Center Sp. z o.o., Kobylniki
  - Szpital Wojewdzki w Koszalinie im. Mikoaja Kopernika, Koszalin
  - University Hospital, Krakow
  - Szpital Kliniczny Nr Pozna?, Poznan
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie w Warszawie, Warsaw
  - Dolnoslaskie Centrum Onkologii - Lower Silesian Oncology Center, Wroclaw
- Russia (5):
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Hertzen Moscow Oncology Research Center, Moscow
  - Institution of the Russian Academy of Medical Sciences Russian Oncological Research Center n.a. N.N. Blokhin, Moscow
  - Budgetary Healthcare Institution of Omsk Region - Clinical Oncological Dispensary, Omsk
  - Bashkortostan Republican Clinical Oncology Dispensary, Ufa
- South Korea (7):
  - National Cancer Center, Goyang
  - CHA Bundang Medical Center CHA University, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (12):
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital del Mar, Barcelona
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital Universitari Parc Tauli, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Instituto Catalán de Oncología - Hospital Universitario Dr. Josep Trueta, Girona
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital General Universitario Gregorio Marano, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Fundacion Instituto Valenciano de Oncologia IVO, Valencia
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Tungs Taichung Metro Harbor Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital NTUH, Taipei
  - Chang Gung Memorial Hospital CGMH - Linkou Branch, Taoyuan District
- United Kingdom (5):
  - Imperial College Healthcare NHS Trust, London
  - Sarah Cannon Research Institute UK, London
  - University College London Hospital, London
  - Genesis Cancer Care-CHURCHILL Hospital Headington, Oxford
  - Royal Marsden Hospital, Sutton